CLINICAL TRIAL: NCT06237127
Title: Effects of Goji Berry Intake on Risk of Age-related Macular Degeneration: A Randomized Clinical Trial
Brief Title: Effects of Goji vs. Fiber on Macular Degeneration
Acronym: GOJI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Robert Hackman, PhD, Research Nutritionist, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2082960
Record Dates: First submitted 2024-01-19; First posted 2024-02-01 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Age-Related Macular Degeneration
Keywords: Goji Berry; Age-Related Macular Degeneration; Lutein; Zeaxanthin; Fiber; Carotenoids; Gut Microbiome; HDL; Cholesterol Efflux Capacity; Eye Health
MeSH Terms: conditions — Macular Degeneration | interventions — Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Goji berry (Experimental): For the goji berry arm, participants will consume goji berries.
  Interventions: Dietary Supplement: Goji berry
- Fiber (Active Comparator): For the fiber arm, participants will consume fiber supplements that closely matches the fiber type and amount found in the portion of goji berries.
  Interventions: Dietary Supplement: Fiber

INTERVENTIONS:
Dietary Supplement: Goji berry — Participants will be instructed to consume 14 grams of goji berries 5 days a week for 6 months
  Arms: Goji berry
Dietary Supplement: Fiber — Participants will be instructed to consume the fiber supplements 5 days a week for 6 months
  Arms: Fiber

SUMMARY:
The goal of this project is to conduct a clinical trial in 60 participants ranging from age 65-95 who are at risk for age-related macular degeneration (AMD). The study will evaluate the effects of 14g of goji berry intake or an equivalent amount and type of fiber, five days a week for six months, on visual health, gut microbiome profiles, skin carotenoid measures, and lipoprotein profiles.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the third leading cause of blindness worldwide. The disease occurs when the macula in the central retina develops lesions due, in part, to the loss of the protection of macular pigments zeaxanthin, lutein, and meso-zeaxanthin, which are responsible for light filtering and oxidative defense. The major risk factor for AMD is aging, and currently, no definitive prevention for AMD exists.

Goji berry (Lycium Barbarum) is a fruit that has been used as traditional medicine in Asian countries for more than 2,000 years. Modern science has identified potential benefits of the berry in oxidant defense, immune regulation, diabetes, and vision in animal and cell models. Nonetheless, evidence regarding the effects of goji berries on human health is scarce. The bioactive components of goji berries include zeaxanthin, lutein, Lycium Barbarum polysaccharides-protein complex, betaine, cerebroside, minerals, and vitamins. Importantly, goji berries contain the highest concentration of zeaxanthin among all commonly consumed foods.

Previous clinical studies have shown that goji berries have a high bioavailability of zeaxanthin, and that macular pigment optical density (MPOD) was increased after supplementation. This study uses macular pigment optical volume (MPOV; a measure that integrates MPOD across multiple macular eccentricities) as the primary outcome measure. It is unknown if the changes in MPOV will be associated with other functional changes or anatomic conditions in the eye among a population with small drusen, a risk factor for AMD. In addition, the impact of goji berry intake on the gut microbiome profile and associated metabolites is unknown, and potentially important in understanding the mechanism(s) of action.

Participants who meet the eligibility criteria will be enrolled and will be randomized 1:1 to the goji berry arm or fiber arm of the study. Over the course of approximately 180 days, participants will consume the assigned food item five days per week and attend three study visits.

Study visits will include ophthalmic imaging and testing, skin carotenoid measurements, completion of a food record, height, weight, handgrip strength, blood pressure measurement, and fasting blood collection. At 2 timepoints participants will be asked to provide a stool sample (collected within 24 hours of visit).

ELIGIBILITY:
Inclusion Criteria:

* Family history of AMD
* Hyperlipidemia or managed diabetes
* 65 - 95 years of age

Exclusion Criteria:

* Dislike of, or allergy to, goji berries or any of the ingredients in the fiber-rich wafers and gummies (wheat, corn, oats, soy, natural orange flavor, xylitol, annatto, pectin, or other food ingredients)
* Consumption of > 2 alcoholic drinks per day
* Indications of substance or alcohol abuse
* Current or planned use of a blood thinner (e.g., Coumadin, Warfarin) at any time during study
* Use of multi-vitamin or any other supplements that contain lutein and/or zeaxanthin (if willing to stop the supplement, subject can be enrolled 6 months from stop date)
* Taking any new medications started within the past 6 months, or changes in medication regimen planned in the next 6 months (stable use greater than 6 months is not exclusionary)
* Any planned international travel during the study
* Consuming >3 servings/day of a combination of spinach, kale, lettuce, orange bell peppers, corn, parsley, squash, broccoli, pumpkin, edamame
* Regularly consuming >3 eggs/day
* Currently participating in any other interventional research study
* Diagnosed with inflammatory bowel disease, irritable bowel syndrome, other gastrointestinal disorder, undergoing cancer therapy or immunocompromised, or diagnosis of another condition where lutein, zeaxanthin and/or fiber supplementation would be contraindicated or would interfere with ability to participate in the study
* Any physical characteristic or condition that precludes ability to perform study procedures
* Medical or psychiatric condition that, in the opinion of the Investigator, would compromise study findings or prevent the participant from completing the study

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Macular pigment optical volume (MPOV) | Day 0 and Day 180
  MPOV provides an objective measure of macular pigments by using dual wavelength autofluorescence using the Heidelberg Spectralis to obtain HRA + OCT measures

SECONDARY OUTCOMES:
Stool microbiome | Day 0 and Day 180
  Metagenomic sequencing
Spectral Domain-Ocular Coherence Tomography (SD-OCT) | Day 0 and Day 180
  Central subfield thickness will be measured using the OCT instrument's algorithm
Fundus autofluorescence (FAF) | Day 0 and Day 180
  Blue FAF imaging will be performed to assess variations in lipofuscin autofluorescence
Color Fundus Photography (CFP) | Day 0 and Day 180
  CFP imaging uses a standard retinal camera.
Microperimetry testing | Day 0 and Day 180
  Microperimetry will be tested according to a standard protocol using a Nidek MP-1 instrument
Dark adaptometry | Day 0 and Day 180
  Dark adaptometry will be assessed using a standard protocol.
Plasma microbial metabolites | Day 0 and Day 180
  Biogenic amines will be measures by LC-MS
Plasma lutein and zeaxanthin | Day 0 and Day 180
  Plasma concentrations of lutein and zeaxanthin will be measured by LC-MS
Lipoprotein profile | Day 0 and Day 180
  Lipoprotein profiles will be measured according to standard protocols
HDL particle characteristics | Day 0 and Day 180
  Plasma will also be used to isolate and characterize HDL particles.
Peripheral blood mononuclear cells (PBMC) gene expression changes | Day 0 and Day 180
  PBMCs will be collected to monitor gene expression changes.
Cognitive function | Day 0 and Day 180
  Cognitive function will be assessed using web-based CANTAB tests
Handgrip strength | Day 0 and Day 180
  Handgrip strength will be measured using a Jamar hand dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Hackman, PhD, Principal Investigator — University of California, Davis; Angela M Zivkovic, PhD, Principal Investigator — University of California, Davis; Glenn Yiu, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Eye Center, Tschannen Eye Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No